CLINICAL TRIAL: NCT05165069
Title: The Efficacy and Safety of Mecobalamin in the Prevention of Capecitabine Induced Hand Foot Syndrome in Breast Cancer Patients: A Multicenter, Phase III, Randomized, Double-blind, Controlled Trial
Brief Title: The Efficacy and Safety of Mecobalamin in the Prevention of Capecitabine Induced Hand Foot Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-KY-007
Record Dates: First submitted 2021-12-15; First posted 2021-12-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hand-foot Syndrome
Keywords: Hand-foot Syndrome, Mecobalamin, Capecitabine, Breast Cancer
MeSH Terms: conditions — Hand-Foot Syndrome; Breast Neoplasms | interventions — mecobalamin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mecobalamin group (Experimental): Mecobalamin (0.5mg / time, 3 times / day) for 6 months
  Interventions: Drug: Mecobalamin 5 MG Disintegrating Oral Tablet
- Placebo group (Placebo Comparator): placebo (0.5mg / time, 3 times / day) for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mecobalamin 5 MG Disintegrating Oral Tablet — Mecobalamin 0.5mg / time, 3 times / day,was taken continuously for 6 months
  Arms: Mecobalamin group
Drug: placebo — placebo 0.5mg / time, 3 times / day,was taken continuously for 6 months
  Arms: Placebo group

SUMMARY:
A multicenter, randomized, placebo-controlled, double-blind, phase III clinical trial will be conducted to explore the efficacy and safety of mecobalamin in the prevention of 2/3 HFS in patients with early breast cancer. 234 patients will be enrolled and will be randomized into mecobalamin group and placebo group at the ration of 1:1. The incidence of grade 2 / 3 HFS in the experimental group and the control group will be observed. This study is expected to provide evidence for clinical prevention of hand foot syndrome, improve clinical treatment guidelines for early breast cancer, and provide reference for other antitumor drugs for hand foot syndrome.

DETAILED DESCRIPTION:
Capecitabine is a drug recommended for adjuvant therapy in early breast cancer. The key to improving the prognosis of early breast cancer is to ensure that adequate treatment is sufficient. Hand foot syndrome Hand foot syndrome (HFS) is the most common and specific side effect of capecitabine, in which the incidence of grade 2 / 3 HFS requiring treatment is as high as 17-36%. At present, there is no specific drug for the treatment of HFS, and capecitabine must be reduced or stopped in case of grade 2 / 3 HFS. The guidelines also do not recommend standard drugs for the prevention of HFS. Mecobalamin is a derivative of vitamin B12, which can improve autonomic nervous system After symptoms and repair of small neuropathy, its clinical indication is the treatment of peripheral neuropathy.

A multicenter, randomized, placebo-controlled, double-blind, phase III clinical trial will be conducted to explore the efficacy and safety of mecobalamin in the prevention of 2/3 HFS in patients with early breast cancer. 234 patients will be enrolled and will be randomized into mecobalamin group and placebo group at the ration of 1:1. The incidence of grade 2 / 3 HFS in the experimental group and the control group will be observed. This study is expected to provide evidence for clinical prevention of hand foot syndrome, improve clinical treatment guidelines for early breast cancer, and provide reference for other antitumor drugs for hand foot syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18 to 75
2. Her-2 negative patients with non metastatic breast cancer.
3. patients with early breast cancer who did not receive PCR after neoadjuvant chemotherapy or patients with lymph node metastasis after breast cancer surgery.
4. Prepare to receive postoperative adjuvant single drug capecitabine or capecitabine combined with endocrine therapy and / or radiotherapy

   The Binbin dose is 1000mg / ㎡, bid (continuous oral administration for 14 days, stopping for 7 days, repeated every 21 days)
5. Eastern cancer cooperation group (ECoG) physical strength score 0-1;
6. During randomization, the toxicity related to previous treatment must be alleviated to NCI CTCAE (version 4.03) ≤ 1 degree (except hair loss or according to the research)

   Other toxicity judged by the investigator that there is no risk to the safety of the patient);
7. Blood routine examination was basically normal within 4 weeks before enrollment: A. white blood cell count (WBC) ≥ 3.0 × 10 ^ 9 / L, B. medium

   Sex granulocyte count (ANC) ≥ 1.5 × 10 ^ 9 / L, C. platelet count (PLT) ≥ 100 × 10^9／L;
8. The liver and kidney function tests were basically normal within 4 weeks before enrollment (based on the normal values in the laboratories of each research center): a

   Total bilirubin (TBIL) ≤ 1.5 × Upper limit of normal value (ULN), B. alanine aminotransferase and aspartate aminotransferase (ALT / AST)

   ≤2.5 × ULN (patients with liver metastasis) ≤ 5 × ULN), C. serum creatinine ≤ 1.5 × ULN or creatinine clearance (CCR)

   ≥60 ml/min；
9. Women of childbearing age must have a serum / urine pregnancy test 4 weeks before enrollment, and the result is negative, and are willing to participate in the study

   Use a medically recognized high-efficiency contraceptive during and within 6 months after the last administration of the drug;
10. Informed consent has been signed before joining the group;
11. There was no active infectious disease within 12 weeks of screening period

Exclusion Criteria:

1. in the first 5 years of randomised allocation, there was a history of malignancy except for breast cancer, but the risk of metastasis or death was negligible.

   Except for malignant tumors that can be cured after treatment (such as appropriately treated cervical carcinoma in situ, non melanoma skin cancer or stage I cancer)

   Uterine cancer, thyroid cancer, etc.);
2. Any accompanying disease or condition that may interfere with the study, or any serious medical impairment that may affect the safety of the subject

   (for example, uncontrollable heart disease, hypertension, active or uncontrollable infection, active hepatitis B virus infection);
3. there are diseases affecting skin: diabetes, dermatomyositis, sclerosing disease, lupus erythematosus and so on.
4. Known history of psychotropic substance abuse or drug abuse;
5. Pregnant or lactating patients;
6. Inability to swallow, intestinal obstruction or other factors affecting drug administration and absorption.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 2 / 3 hand foot syndrome | 6 months
  The incidence equals the numbers of patients happens 2nd or 3rd level hand foot syndrome/the number of total patients in each group

SECONDARY OUTCOMES:
The reduction or withdrawal rate of capecitabine | 6 months
  the proportion of subjects with capecitabine reduction of more than 75% or capecitabine withdrawal accounted for the proportion of subjects in each group
Disease Free Survival | 5 years
  The time from the beginning of treatment to the recurrence of the disease or death from any cause or the end of the visit
Overall Survival | 5 year
  The time from the beginning of treatment to the death of the patient caused by any factor
The score of life quality questionnaire | 6 months
  The score of HF-Qol
The score of life quality | 6 months
  The score of QLQ-C30
The score of life quality QLQ-BR23 | 6 months
  The score of QLQ-BR23
The incidence of adverse events | 6 months
  Incidence of adverse outcome events (such as fatigue, malignancy / vomiting, abdominal pain, diarrhea, stomatitis, impaired liver function, bone marrow suppression, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gong, Study Chair — Sun Yat-sen Memorial Hospital of Sun Yat-sen Univeristy
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xia Y, Zhu Y, Ling L, Xu F, Yang Y, Ye J, Tan W, Chen Z, Liu Q, Wei W, Zhang J, Zhang A, Zhang L, Song E, Gong C. Effect of methylcobalamin on capecitabine induced hand-foot syndrome in patients with HER2 negative early breast cancer: multicentre, double blind, randomised, placebo controlled, phase 3 trial. BMJ. 2025 Sep 11;390:e084290. doi: 10.1136/bmj-2025-084290. PMID 40935571